CLINICAL TRIAL: NCT00096369
Title: An Exploratory Study to Identify Potential Surrogate Endpoint Biomarkers That Are Modulated by Tamoxifen vs. Placebo in Women With an Increased Risk for Breast Cancer
Brief Title: Tamoxifen in Preventing Breast Cancer in Women at Increased Risk for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual goal not met
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000393444; V-10604
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; lobular breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of tamoxifen may be effective in preventing breast cancer.

PURPOSE: This randomized phase II trial is studying tamoxifen to see how well it works compared to placebo in preventing breast cancer in women who are at increased risk for the disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare molecular markers of proliferation and apoptosis in breast epithelial tissue of women at increased risk for breast cancer treated with tamoxifen vs placebo.
* Compare the modulation of markers of genomic instability in breast epithelial tissue of patients treated with these drugs.
* Compare serum levels of IGF-1, IGF-2, and IGFBP-3 of these patients at baseline and after treatment with these drugs.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to estimated 5-year breast cancer risk (1.67-5% vs ≥ 5%), presence of atypical ductal hyperplasia (yes vs no), and menopausal status (premenopausal vs postmenopausal). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral tamoxifen once daily.
* Arm I: Patients receive oral placebo once daily. Treatment in both arms continues for 3 months in the absence of invasive breast cancer or unacceptable toxicity.

Patients undergo core needle biopsy and fine needle aspiration biopsy at baseline and then at the completion of study treatment (for premenopausal patients); exactly 84 days after the first biopsy (for postmenopausal patients); or on the first or second day of the menstrual cycle on or after 84 days (during the third menstrual cycle) after the first dose of study medication (for patients with irregular menses).

Patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 130 patients (65 per arm) will be accrued for this study within 30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk for breast cancer, as defined by 1 of the following criteria:

  * Histologically confirmed lobular carcinoma in situ (LCIS) treated by local excision only
  * Composite increased breast cancer risk of ≥ 1.67% over 5 years, based on the following criteria:

    * Age
    * Number of first-degree female relatives with breast cancer
    * One or more prior breast biopsies

      * Fine-needle aspiration cytology of a non-cystic lesion in lieu of an open biopsy is considered a biopsy
    * Prior diagnosis of atypical hyperplasia of the breast
    * Age at first live birth
    * Nulliparity
    * Race
    * Age at onset of menarche
* No prior or suspected invasive breast cancer or ductal carcinoma in situ
* No clinical evidence of malignancy by physical examination, including a breast examination within the past 3 months
* No evidence of suspicious or malignant disease or uncharacterized lesions on bilateral mammogram within the past 6 months
* Normal gynecologic examination, including a bimanual pelvic examination and, if indicated, pap smear within the past 12 months
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 35 and over

Sex

* Female

Menopausal status

* Premenopausal and ovulating*, defined as having regular menses for the past 6 months OR irregular menses with follicular phase (i.e., day 3) follicle-stimulating hormone level < 20 mIU/mL OR
* Postmenopausal NOTE: * Ovulation is determined by day 21 progesterone level > 3 ng/mL

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Complete blood count normal
* No active bleeding disorder (e.g., qualitative or quantitative platelet abnormality, hemophilia, or von Willebrand's disease)

Hepatic

* Liver function tests normal

Renal

* Not specified

Cardiovascular

* No prior deep-vein thrombosis except a single occurrence related to lower extremity trauma
* No prior cerebral vascular accident
* No prior transient ischemic attack

Pulmonary

* No prior pulmonary embolus except a single occurrence related to lower extremity trauma

Other

* No saline or silicone breast implants
* No known allergy to tamoxifen
* No macular degeneration
* No malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No nonmalignant disease that would preclude administration of tamoxifen
* No psychiatric condition, including a history of clinical depression or addictive disorder, that would preclude giving informed consent or study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic adjuvant chemotherapy for LCIS

Endocrine therapy

* No prior tamoxifen, raloxifene, or other selective estrogen-receptor modulators
* At least 3 months since prior and no concurrent use of any of the following drugs:

  * Estrogen or progesterone replacement therapy
  * Oral contraceptives
  * Androgens
  * Luteinizing hormone-releasing hormone analogs
  * Prolactin inhibitors
  * Antiandrogens
  * Steroids
* No concurrent steroids for asthma

Radiotherapy

* No prior radiotherapy for LCIS

Surgery

* No prior bilateral prophylactic mastectomy
* No prior mastectomy for LCIS

Other

* Concurrent nonhormonal medications allowed
* No concurrent warfarin or cholestyramine
* No prior or concurrent participation in any other cancer prevention study

  * Patients treated with placebo on protocol NSABP-P-1 are eligible

Ages: 35 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2000-02 (Actual); Primary Completion 2007-03-15 (Actual); Study Completion 2007-03-15 (Actual)

PRIMARY OUTCOMES:
Plasma levels of hormones and binding proteins as measured by ELISA, IHC, and TUNEL at baseline and 3 months
Markers of proliferation and apoptosis in breast cells as measured by quantitative MSP at baseline and 3 months
Promoter-region methylation as assessed by microarrays at baseline and 3 months
Gene expression

CONTACTS AND LOCATIONS:
Overall Officials: David M. Euhus, MD, Principal Investigator — Simmons Cancer Center
Locations (4):
- United States (4):
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas